CLINICAL TRIAL: NCT00592241
Title: Self Operating of the ADI Insulin Pump By Intended Users - A Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NiliMedix (Industry)
Responsible Party: Dr. Hanna Levy, Clinical Study Consultant, NiliMedix
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: NM-UA-01
Record Dates: First submitted 2007-12-17; First posted 2008-01-14 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus
Keywords: Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (No Intervention): Subject is diagnosed as a diabetic, or subject is parent/guardian of a diabetic child age under 18 years.
  Interventions: Device: "Adi" Insulin Pump Usability

INTERVENTIONS:
Device: "Adi" Insulin Pump Usability — no intervention
  Other Names: "Adi" Insulin Pump

SUMMARY:
Diabetes mellitus (DM) is a multisystem disease with both biochemical and anatomical consequences. Insulin pump therapy (continuous subcutaneous insulin infusion [CSII]) is an attractive way of treating patients with diabetes. The NiliMedix ADI Insulin Pump is an ambulatory, battery operated, rate programmable micro infusion pump, designed for continuous delivery of insulin.

Insulin pumps require extensive user interaction because it is critical for treatment. Avoidance of use-related risks that could harm the patient or impact the quality of the treatment is important. Testing for ease and accuracy of use is the only way to ensure that users can safely and effectively operate, install, and program and maintain the insulin pump device.

DETAILED DESCRIPTION:
This usability study was designed in order to test independent home use and device interface effectiveness of the NiliMedix Adi Insulin Pump, in order to validate safe and effective use by intended users. The study objectives are as following:

* Validate the safe and effective use while using the ADI Insulin Pump by intended users. This objective will be assessed by carrying out list of tasks (operating the device, programming the appropriate flow rate and volume-to-be-infused parameters, and reacting to hazard massages) independently and successfully.
* Evaluate user's satisfaction. Study Design Orientation, consent, and pre-test questionnaire Participants will receive a short, scripted verbal orientation explaining the purpose of the usability test.

Prior to any study related procedures participant will provide written informed consent.

Performance evaluation The performance evaluation will consist of a list of tasks that participants will attempt to complete. The tasks were designed to explore the usability concerns. Participants will be provided with the Adi Insulin Pump and the user manual.

All participants will be guided by the investigator how to use the ADI Insulin Pump independently, how to read and interpret the display readings, how to program the device including insulin Basal and Bolus settings as well as how to maintain the device. In addition, participants will be given sufficient time to read carefully the user manual.

After ensuring that the participant has perceived the directions for use he will be asked to operate the Adi Insulin Pump by performing list of tasks.

All tasks will be conducted by the participants independently. The investigator will not guide the subject during this phase- unless the subject asked him to.

ELIGIBILITY:
Inclusion Criteria:

* Male/female age 18 years and up.
* Subject is diagnosed as a diabetic, or subject is parent/guardian of a diabetic child age under 18 years.
* Subject understands the study procedure.
* Subject is able to read the User Manual.
* Signed Informed Consent form
* Compliance with study requirements.

Exclusion Criteria:

* Major physical, motor, mental, behavioral, or psychiatric limitations.
* Concurrent additional major illness.
* Subject objects to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Validate safety while using the ADI Insulin Pump by intended users. This objective will be assessed by independently and successfully carrying out a list of tasks. | 4 hours

SECONDARY OUTCOMES:
Evaluate user's satisfaction. | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Naim Shehadah, Prof., Principal Investigator — RAMBAM Medical Center, Haifa Israel
Locations (1):
- RAMBAM Medical center, Haifa, Israel